CLINICAL TRIAL: NCT00230841
Title: Efficacy of Optimal Versus 'Traditional' Delivery of Humidity in Children With Croup
Brief Title: Comparing Different Ways of Delivering Humidity to Children With Croup
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Collaborators: The Physicians' Services Incorporated Foundation (Other)
Responsible Party: Principal Investigator, Dennis Scolnik, Staff Physician, The Hospital for Sick Children
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0020010158
Record Dates: First submitted 2005-09-29; First posted 2005-10-03 (Estimated); Last update posted 2013-08-02 (Estimated); Status verified 2013-07

CONDITIONS: Croup
Keywords: croup; humidity therapy; pediatrics
MeSH Terms: conditions — Croup

INTERVENTIONS:
Device: nebulized humidity

SUMMARY:
Croup affects 5% of children under 6 years of age, resulting in visits to hospital Emergency Departments, and in 1% of children, hospitalization. Traditionally, the first therapy offered is humidification which can liquify airway secretions and decrease airway swelling. This study will compare the effectivenesss of 40% and 100% humidity through a specially designed machine called a nebulizer, with the usual humidity set-up (blown into the patient's face from a hose).

ELIGIBILITY:
Inclusion Criteria:

* children aged 3 months - 10 years
* croup score greater than or equal to 2 after a 30 minute waiting period

Exclusion Criteria:

* Symptoms of croup requiring immediate intervention with nebulized epinephrine or intubation
* symptoms or signs of alternative causes of stridor
* inability of caregivers to understand or speak English and/or sign for informed consent
* history of chronic pulmonary disease except for asthma, or co-existent systemic disease
* previous history of intubation
* duration of present illness >1 week
* systemic or inhaled glucocorticoids in previous 48 hours
* epinephrine in previous 4 hours

Ages: 3 Months to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 129
Dates: Start 2001-09; Study Completion 2004-04

PRIMARY OUTCOMES:
changes in the croup score from baseline to 30 and 60 minutes

SECONDARY OUTCOMES:
steroid or epinephrine treatment at 60 minutes
discharge rate at 60 minutes
change in pulse, respiratory rate, and oxygen saturation at 60 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Dennis Scolnik, MD, Principal Investigator — The Hospital for Sick Children, Toronto Canada
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada

REFERENCES:
- [Result] Scolnik D, Coates AL, Stephens D, Da Silva Z, Lavine E, Schuh S. Controlled delivery of high vs low humidity vs mist therapy for croup in emergency departments: a randomized controlled trial. JAMA. 2006 Mar 15;295(11):1274-80. doi: 10.1001/jama.295.11.1274. PMID 16537737